CLINICAL TRIAL: NCT06611072
Title: OveRcoming immunosupprEssion aNd rebAlancing the Immune reSponSe in ovAriaN CancEr Study
Acronym: RENAISSANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gynaecologisch Oncologisch Centrum Zuid (Other)
Collaborators: Eindhoven University of Technology (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jurgen M.J. Piek, MD, PhD, Gynaecologisch Oncologisch Centrum Zuid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL8439200023
Record Dates: First submitted 2024-08-04; First posted 2024-09-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer; Ovarian Carcinoma; Immune Suppression; Immune System Suppression
Keywords: Ovarian cancer; Immune system; Immune suppression; Immune system suppression; Immunotherapy; Monocytes; Myeloid cells; Vena punction; Bone marrow aspiration; Spleen biopsy; Peritoneal fluid; Tumor biopsy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: investigator-initiated, multi-center explorative cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Patients with OC who undergo primary debulking surgery
  Interventions: Procedure: Bone marrow aspiration; Procedure: Vena puncture; Procedure: Peritoneal fluid; Procedure: Spleen biopsy; Procedure: Tumor biopsy; Procedure: Omental biopsy
- Group 2 (Experimental): Patients with OC who undergo interval debulking surgery
  Interventions: Procedure: Bone marrow aspiration; Procedure: Vena puncture; Procedure: Peritoneal fluid; Procedure: Spleen biopsy; Procedure: Tumor biopsy; Procedure: Omental biopsy
- Group 3 (Active Comparator): Controls as blood and bone marrow donors
  Interventions: Procedure: Bone marrow aspiration; Procedure: Vena puncture; Procedure: Peritoneal fluid

INTERVENTIONS:
Procedure: Bone marrow aspiration — Bone marrow samples will be obtained from the sternum or the iliac crest according to standard practice by experienced operators during the surgery patients will undergo as part of their medical treatment. BM mononuclear cells will be isolated using Ficoll-Paque and progenitor cells will be enriched using positive selection with CD34 beads by MACS. Progenitor cell composition will be identified using flow cytometry. HSPC proliferation assays (standard CFU assays) to assess myeloid colony-forming potential will be performed. In addition, single-cell RNA- sequencing and epigenetic assessment (ATAC-seq, ChIP-seq, DNA methylation) will be performed.
Procedure: Vena puncture — Whole blood will be collected and peripheral blood mononuclear cells (PBMC) will be isolated using Ficoll-Paque. Cellular subpopulations will be purified using negative selection of monocytes with PanMonocyte beads by MACS.
Procedure: Peritoneal fluid — Peritoneal fluid will be collected during the surgery.
Procedure: Spleen biopsy — Spleen samples will be obtained by experienced surgeons during the debulking surgery. Spleen mononuclear cells will be isolated using Ficoll-Paque and progenitor cells will be enriched using positive selection with CD34 beads by MACS. Cellular subpopulations will be further purified using negative selection of monocytes with PanMonocyte beads by MACS. Progenitor cell composition will be identified using flow cytometry. HSPC proliferation assays (standard CFU assays) to assess myeloid colony-forming potential will be performed. In addition, single- cell RNA-sequencing and epigenetic assessment (ATAC-seq, ChIP-seq, DNA methylation) will be performed.
  Arms: Group 1; Group 2
Procedure: Tumor biopsy — During debulking surgery, all visible tumor tissue will be removed by experienced surgeons.
  Arms: Group 1; Group 2
Procedure: Omental biopsy — During debulking surgery, an omental biopsy will be done.
  Arms: Group 1; Group 2

SUMMARY:
Ovarian cancer (OC) is one of the most lethal cancers in the world due to late-stage disease at diagnosis. Standard therapy consists of debulking surgery and chemotherapy. However, despite this aggressive treatment, recurrent disease almost invariably occurs resulting in a five-year survival rate of approximately 30%.

Immunotherapy could be a way to increase survival in OC patients. However, a major barrier to a successful deployment of cancer immunotherapy for ovarian cancer patients is the immunosuppressive tumor microenvironment.

Envisioned solution/research direction

Tumor-related inflammation is one of the hallmarks of cancers in general. Innate immunity specifically is a common denominator that is involved in the pathogenesis of OC. To improve the patient's outcome and identify novel therapeutic targets, one needs a deeper understanding of the tumor-induced changes in the bone marrow myeloid progenitor cells. Furthermore, treatment of these cells by nanoparticles or other agents that induce a program of 'trained immunity' may be a novel way to re- educate myeloid cells and their bone marrow progenitors in OC patients.

Hypothesis

We hypothesize that by exposing myeloid cells or their progenitors to various agents that induce trained immunity (e.g. trained immunity-inducing agents: BCG, heat-killed Candida,), these immune cells will undergo functional reprogramming to induce a tumor-suppressive phenotype. In the future, this could be explored as a novel immunotherapy for tumors that are refractory to conventional treatment.

Objective

To characterize and phenotype the immune state of OC patients compared to controls without cancer with a focus on the hematopoietic organs and the immune cells originating from these organs. In addition, the effect of established trained immunity-inducing agents on these cells will be evaluated in vitro, potentially providing new therapies.

This will be executed by assessing the transcriptional, epigenetic, and functional reprogramming of circulating monocytes and myeloid progenitor cells in OC and by assessing the in vitro effect of trained immunity inducers on the reprogramming of circulating monocytes and myeloid progenitor cells.

Study design: investigator-initiated, multi-center explorative cross-sectional study at the Catharina hospital Eindhoven, Radboud University Medical Center and Eindhoven University of Technology.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Problem description/ unmet needs:

Ovarian cancer is the fifth leading cause of cancer death among women in the Western world. The high mortality rate is due to detection at an advanced stage of the disease and lack of curative therapies. Standard therapy consists of a combination of cytoreductive surgery and chemotherapy. Despite this aggressive treatment, recurrent disease almost invariably occurs resulting in a five-year survival rate of only 30%, which has not changed significantly over the last 30 years.

Recurrent ovarian cancer is generally treated with second/third line chemotherapy, and (costly) targeted therapies. Although targeted therapy options are rapidly expanding, response rates often fall short of expectations probably caused by heterogeneity of the disease. Therefore, new treatment options need to be explored. One such option is immunotherapy. However, the limited data on this topic show disappointing results.

Envisioned solution/research direction:

To improve the patients' outcomes and identify novel therapeutic targets, one needs a 'systems understanding' of the pathophysiology of tumors, which transcends beyond the process of carcinogenesis to encompass the complex interaction of the malignant cells with other cell types in the tumor and the tumor environment (TME), especially immune cells. The inflammatory TME has characteristics that promote and support the malignant phenotype, and inflammatory pathways have been proposed as new targets for cancer therapy. The TME conditions the local myeloid cells to become immunosuppressive. In this project we primarily focus on myeloid cells, in particular circulating monocytes and their progenitors, as well as the tumor-

associated macrophages (TAMs) which are pluripotent myeloid cells that represent the most abundant component of the TME in advanced OC arguing for their importance in the pathogenesis of OC.

In the present study, we aim to investigate the programming of myeloid cells in OC patients with advanced tumors in depth and to explore whether we can functionally reprogram myeloid cells from different bodily compartments (circulating monocytes, bone marrow (BM) and spleen progenitors) towards an anti-tumorigenic phenotype by trained immunity-modulating nanoparticles. If this hypothesis is proven to be correct, this mechanism could be explored in further studies including investigation of the interaction of myeloid cells with other immune cells and as a novel immunotherapy for OCs that are refractory to conventional treatment.

OBJECTIVES

To assess the transcriptional, epigenetic, and functional reprogramming of circulating monocytes and myeloid progenitor cells in OC by in vitro exposure to agents that modulate trained immunity.

To achieve this goal the study has a set of complementary key objectives:

To assess the transcriptional, epigenetic, and functional signature of i) circulating monocytes in patients with OC compared to controls in response to trained immunity inducers in vitro and ii) bone marrow and spleen myeloid progenitor cells in patients with OC compared to controls in response to trained immunity inducers in vitro.

STUDY DESIGN

This is an investigator-initiated, single-center cross-sectional explorative study that will be performed in the Catharina hospital Eindhoven at the Department of Obstetrics and Gynecology, Division of gynecological oncology in collaboration with the Eindhoven University of Technology and the department of internal medicine, Radboud UMC.

All OC patients and controls will donate blood samples during the operation. The OC patients will undergo surgery for removal of their tumor (as planned by their treating physician) and will be requested permission to use small samples of their removed tissue (malignant and benign samples), a BM sample from sternum or posterior iliac crest and spleen). The controls will undergo surgery for benign gynecological conditions (as planned by their treating physician) and will be requested permission to use a BM sample from sternum or posterior iliac crest.

The following set of measurements will be performed on peripheral blood samples:

Circulating and splenic monocytes will be purified and the following assessments will be performed before and after treatment with trained immunity inducers:

* Transcriptome analysis by RNA-sequencing
* Epigenetic analysis of chromatin accessibility (ATACseq), whole-genome histone modification profiles, and DNA methylation
* Immunological profiling of the monocytes by stimulation and trained immunity assays

The following set of measurements will be performed on bone marrow aspirates:

Bone marrow and splenic progenitor cells will be purified and the following assessments will be performed before and after treatment with trained immunity- inducing agents:

* Transcriptome analysis by RNA-sequencing
* Epigenetic analysis of accessibility (ATACseq), whole-genome histone modification profiles, and DNA methylation
* Composition, differentiation, and immunological profiling of the progenitors by colony formation, differentiation, stimulation, and trained immunity assays

All experiments and handling of samples will be performed according to Good Clinical Practice and the declaration of Helsinki.

The effect of exposure to trained immunity inducing agents on the functional phenotype of the monocytes and progenitors will be interrogated by pathway analysis of transcriptome and epigenome, to identify the major cellular processes in reprogramming circulating monocytes and progenitors.

STUDY POPULATION

The following patient groups will be included in the study:

Group 1. Patients with OC undergoing primary debulking surgery (N=30) Group 2. Patients with OC undergoing interval debulking surgery (N=30) Group 3. Controls as blood and bone marrow donors (N=30)

Rationale for the choice of study subjects:

Data from controls is crucial in order to provide a baseline, make useful comparisons, and to legitimately analyze immune cell status of OC patients and the effects of trained immunity-inducing agents. Both OC patients who are chemotherapy naïve (primary debulking) and who have had chemotherapy (carboplatin-paclitaxel) will be included in this study, to determine the effect of chemotherapy on the TAMs.

Subject recruitment: controls will be recruited from patients who undergo surgery for benign gynecological conditions. Patients will be invited to participate by their treating gynecologist during an outpatient clinic visit or via a letter. In addition, they will receive a letter with study-related information. Within one week they will be contacted to check if they require additional information and if they are willing to participate.

Patients with OC will be recruited if they undergo debulking surgery at our centers. Patients will be invited to participate by their treating gynecological oncologist during an outpatient clinic visit or via a letter; in addition, they will receive a letter with study-related information. Within one week they will be contacted to check if they require additional information and if they are willing to participate.

Approximately 150 patients undergo surgery for benign gynecological conditions at our department and around 100 patients undergo debulking surgery at our center annually. Therefore, inclusion of the limited number of subjects aimed for this study is feasible within three years.

Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Subjects should be at least 18 years old and mentally competent
* Newly diagnosed patients with OC who go for primary debulking surgery or OC are scheduled for interval debulking
* Controls: women who undergo abdominal surgery for benign gynecological conditions under general anesthesia

Exclusion criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Mentally incompetent
* Pregnant or breastfeeding
* Known inflammatory or infectious diseases or an immunosuppressive status;
* Using medication interfering with the immune system
* Severe comorbidities: other active malignancy (except for basal cell carcinoma and other in situ carcinomas)
* Serious psychiatric pathology
* A self-reported alcohol consumption of >21 units per week

Sample size calculation:

The whole-genome analyses (transcriptome, epigenome) and systems biology models that will be performed during the current study will encompass a very large number of variables, each with different variations within the samples. Therefore, due to the nature of the methodological approach, the calculation of the precise number of samples is not possible. Based on the previous whole-genome transcriptional and epigenetic analyses of human macrophages, we will compare full transcriptional and epigenetic profiles of macrophages and TAMs differentiated from groups of 30 patients who received neoadjuvant chemotherapy and 30 patients who are chemo naïve and 30 patients with benign gynecological disease. The above-mentioned numbers of subjects are determined after careful consideration and shared consensus by members of the scientific team involved in the study. The exploratory nature of the study and, in case of invasive investigations, the risks and burden on participants were taken into account.

TREATMENT OF SUBJECTS Not applicable as the patients will not undergo other treatments within the study than those already planned by their treating physician corresponding to the standard of care.

INVESTIGATIONAL PRODUCT Trained-immunity modulating nanoparticles and cytokines that have shown to induce trained immunity.

NON-INVESTIGATIONAL PRODUCT Not applicable

METHODS

Study parameters/endpoints

Main study parameter/endpoint Transcriptional, epigenetic, and functional signature of circulating monocytes and myeloid progenitors before and after in vitro exposure to trained immunity-modulating nanoparticles and/or trained immunity-inducing cytokines from women with ovarian cancer and controls with benign gynecological disease.

Secondary study parameters/endpoints Not applicable

Other study parameters Besides the above-mentioned parameters, the following parameters will be collected in all patients and controls (if applicable):age, length, weight, treatment received (surgery, medication), result of treatment (complete remission, incomplete biochemical remission, persistent disease), OC tumormarkers, circulating immune cells counts at the time point when blood will be collected, use of medication, imaging results: tumor size, invasion, location of metastases, histological results, date of diagnosis, surgery date/ start date of medication, complications of treatment, duration of follow-up, smoking habits and alcohol intake. These items can all affect the immune status of the patients and therefore need to be analysed for possible correlation(s) with outcome of results from main parameter.

In case of unexpected findings during the laboratory experiments with clinical relevance for the patient, the principal investigator will be informed and he will inform the treating physician, so he/she can inform the patient.

Randomization, blinding, and treatment allocation Not applicable

Study procedures

Methods and techniques:

Myeloid cells collection and stimulation experiments

Myeloid cells will be collected from four compartments:

1. Whole blood will be collected and peripheral blood mononuclear cells (PBMC) will be isolated using Ficoll-Paque.
2. BM samples will be obtained from the sternum or the iliac crest according to standard practice by experienced operators during the surgery patients will undergo as part of their medical treatment. BM mononuclear cells will be isolated using Ficoll-Paque and progenitor cells will be enriched using positive selection with CD34 beads by MACS. Progenitor cell composition will be identified using flow cytometry. HSPC proliferation assays (standard CFU assays) to assess myeloid colony-forming potential will be performed. In addition, single-cell RNA- sequencing and epigenetic assessment (ATAC-seq) will be performed.
3. Spleen samples (only from patients with OC) will be obtained by experienced surgeons during the debulking surgery. Spleen mononuclear cells will be isolated using Ficoll-Paque and progenitor cells will be enriched using positive selection with CD34 beads by MACS.. Progenitor cell composition will be identified using flow cytometry. In addition, single- cell RNA-sequencing and epigenetic assessment (ATAC-seq) will be performed.
4. Peritoneal fluid will be collected and mononuclear cells will be isolated using Ficoll-Paque. Cell composition will be identified using flow cytometry.

The cell processing (ie. isolation of cells from samples) will be performed at the RadboudUMC laboratory. Functional assays (in vitro cultures, ELISA, flow cytometry, sequencing will be performed at the RadboudUMC laboratory site. The purified cell populations (from blood, bone marrow, and spleen) will be cultured, and trained immunity will be induced by agents that have already shown to induce trained immunity and have the potential to be used as therapeutic agents in vivo: Beta-glucan, Lipopolysaccharide, Mifamurtide, Heat-killed Candida and Bacillus Calmette-Guérin (see sheets per molecule).

These in vitro trained immunity experiments are well established and optimized assays and described in detail before. Briefly, the purified cells are cultured in well plates, are then exposed to trained immunity- inducing agents for 24 hours. 6 days after this primary stimulus, the cells are exposed to an unrelated secondary stimulus (LPS or Pam3cys) and after 24 hours the supernatant of the cells and the cells are collected for further analysis.

Proinflammatory cytokines in the supernatant will be measured by ELISA as immune parameters for monocyte cell function and induction of trained immunity.

Proinflammatory cytokines in the supernatant will be measured by ELISA as immune parameters for monocyte cell function and induction of trained immunity.

In addition, epigenetic reprogramming in the monocytes/macrophages will be assessed by ATAC-seq assays since epigenetic rewiring is a fundamental feature of trained immunity.

In order to correctly interpret and analyze the results, it is crucial to compare the trained state of the patients' immune cells to the immune cells of healthy donors. We expect that immune cells from OC patients have a more tolerant (i.e., less trained) immune state compared to controls, as has recently shown to be the case in for example thyroid cancer. We also expect that these cells can be modulated in vitro with the trained immunity- inducing agents, reverting the tolerant state and bringing it to the level of the controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be at least 18 years old and mentally competent;
* Newly diagnosed patients with OC who go for primary debulking surgery or patients with OC who are scheduled for interval debulking;
* Controls: women who undergo surgery for benign gynaecological conditions under general anaesthesia.

Exclusion Criteria:

* Mentally incompetent;
* Pregnant or breastfeeding;
* Known inflammatory of infectious diseases or an immunosuppressive status;
* Using medication interfering with the immune system;
* Severe comorbidities: other active malignancy (except for basal cell carcinoma and other in situ carcinomas);
* Serious psychiatric pathology;
* A self reported alcohol consumption of >21 units per week.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cell composition of immune organs using flow cytometry | 3 years including evaluation phase
  The number and ratios of different types of stem and immune cells will be determined using general cell protein markers in combination with flow cytometry. Analysis will be performed on blood, spleen, bone marrow and the intraperitoneal fluid.
Cell composition and epigenetic status of cells of immune organs using ATAC and RNA sequencing | 3 years including evaluation phase
  Cell ratios and epigenetic profile of immune cells in the blood, tumor, bone marrow, and spleen will be analyzed using single-cell RNA and single-cell ATAC sequencing.
Trained immunity response | 3 years including evaluation phase
  We focus on the degree of trained immunity response upon ex vivo stimulation with trained immunity inducers and measured as the concetration of inflammatory cytokines and ROS production.

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No